CLINICAL TRIAL: NCT05931874
Title: Fit2ThriveMIND: Optimizing a mHealth Physical Activity Intervention With Mindful Awareness Lessons in Breast Cancer Survivors
Brief Title: Optimizing a mHealth Physical Activity Intervention With Mindful Awareness Lessons in Breast Cancer Survivors
Acronym: F2TMind
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Siobhan M Phillips, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: NU 22CC05; R01CA266178 (NIH)
Record Dates: First submitted 2023-05-24; First posted 2023-07-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; e-health; physical activity; mindfulness
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: The four Intervention components that are candidates for inclusion in the optimized intervention, each with 2 possible levels, will be tested in a 24-week intervention with a 24-week follow-up using a MOST approach. The effects of the four individual intervention components and their combinations will be examined via a full factorial experiment. The investigators chose a factorial experimental design because these designs have two characteristics essential to the success of MOST. They: a) separate component effects enabling the estimation of the main effect of each candidate component and interactions between components and b) are more economical compared to alternative designs because they often require substantially fewer subjects to achieve the same power and use less resources. The investigators are using a full factorial experiment with 2^4=16 experimental conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Exp Condition 1 (Experimental): Research participant receives the Core Intervention + E-Coach + General Mindfulness Training + MVPA Specific Mindfulness Training + Buddy
  Interventions: Behavioral: Core Intervention; Behavioral: E-Coach; Behavioral: Buddy; Behavioral: General Mindfulness Training; Behavioral: MVPA-Specific Mindfulness Training
- Exp Condition 2 (Active Comparator): Research participant receives the Core Intervention + E-Coach + General Mindfulness Training + MVPA Specific Mindfulness Training
  Interventions: Behavioral: Core Intervention; Behavioral: E-Coach; Behavioral: General Mindfulness Training; Behavioral: MVPA-Specific Mindfulness Training
- Exp Condition 3 (Active Comparator): Research participant receives the Core Intervention + E-Coach + Buddy
  Interventions: Behavioral: Core Intervention; Behavioral: E-Coach; Behavioral: Buddy
- Exp Condition 4 (Active Comparator): Research participant receives the Core Intervention + E-Coach
  Interventions: Behavioral: Core Intervention; Behavioral: E-Coach
- Exp Condition 5 (Active Comparator): Research participant receives the Core Intervention + E-Coach + General Mindfulness Training + Buddy
  Interventions: Behavioral: Core Intervention; Behavioral: E-Coach; Behavioral: Buddy; Behavioral: General Mindfulness Training
- Exp Condition 6 (Active Comparator): Research participant receives the Core Intervention + E-Coach + General Mindfulness Training
  Interventions: Behavioral: Core Intervention; Behavioral: E-Coach; Behavioral: General Mindfulness Training
- Exp Condition 7 (Active Comparator): Research participant receives the Core Intervention + E-Coach + MVPA Specific Mindfulness Training + Buddy
  Interventions: Behavioral: Core Intervention; Behavioral: E-Coach; Behavioral: Buddy; Behavioral: MVPA-Specific Mindfulness Training
- Exp Condition 8 (Active Comparator): Research participant receives the Core Intervention + E-Coach + MVPA Specific Mindfulness Training
  Interventions: Behavioral: Core Intervention; Behavioral: E-Coach; Behavioral: MVPA-Specific Mindfulness Training
- Exp Condition 9 (Active Comparator): Research participant receives the Core Intervention + General Mindfulness Training + Buddy
  Interventions: Behavioral: Core Intervention; Behavioral: Buddy; Behavioral: General Mindfulness Training
- Exp Condition 10 (Active Comparator): Research participant receives the Core Intervention + General Mindfulness Training
  Interventions: Behavioral: Core Intervention; Behavioral: General Mindfulness Training
- Exp Condition 11 (Active Comparator): Research participant receives the Core Intervention + MVPA Specific Mindfulness Training + Buddy
  Interventions: Behavioral: Core Intervention; Behavioral: Buddy; Behavioral: MVPA-Specific Mindfulness Training
- Exp Condition 12 (Active Comparator): Research participant receives the Core Intervention + MVPA Specific Mindfulness Training
  Interventions: Behavioral: Core Intervention; Behavioral: MVPA-Specific Mindfulness Training
- Exp Condition 13 (Active Comparator): Research participant receives the Core Intervention + General Mindfulness Training + MVPA Specific Mindfulness Training + Buddy
  Interventions: Behavioral: Core Intervention; Behavioral: Buddy; Behavioral: General Mindfulness Training; Behavioral: MVPA-Specific Mindfulness Training
- Exp Condition 14 (Active Comparator): Research participant receives the Core Intervention + General Mindfulness Training + MVPA Specific Mindfulness Training
  Interventions: Behavioral: Core Intervention; Behavioral: General Mindfulness Training; Behavioral: MVPA-Specific Mindfulness Training
- Exp Condition 15 (Active Comparator): Research participant receives the Core Intervention + Buddy
  Interventions: Behavioral: Core Intervention; Behavioral: Buddy
- Exp Condition 16 (Active Comparator): Research participant receives the Core Intervention
  Interventions: Behavioral: Core Intervention

INTERVENTIONS:
Behavioral: Core Intervention — All participants will receive a low-resource self-monitoring intervention consisting of the Fitbit Alta HR (or similar) and the study self-monitoring app.
  Participants will be provided with the Fitbit Alta HR. They will be asked to download the Fitbit app and wear the Fitbit 24/7 throughout the study. The Fitbit measures PA intensity, steps, and heart rate, and it syncs directly with the Ftibit app on the smartphone which will ill automatically sync with the study app and provide Fitbit data to the study team in real-time.
  The core study app will support BCS to increase their MVPA. The app will also contain educational information on MVPA and effective behavior change strategies for building self-efficacy, overcoming barriers, enhancing facilitators, setting realistic outcome expectations, and self-regulatory skill-building (i.e., reviewing progress, goal setting, action-planning and coping with disruptions).
Behavioral: E-Coach — Participants assigned to this condition will receive a weekly scheduled text message from their coach. Text messages will focus on building self-efficacy and self-regulation skills, setting realistic outcome expectations, overcoming barriers, and problem-solving and will directly support the participant's engagement in the intervention. The coach will provide a brief overview of the participant's recent progress and goals, ask if they are having any barriers and help them troubleshoot and set specific goals for the next week. Text message protocols will be informed by the investigators' previous experience using telephone coaching to promote MVPA in cancer survivors. In addition to the scheduled messaging, participants will also be instructed to reach out to their coach with any questions or for additional assistance.
  Arms: Exp Condition 1; Exp Condition 2; Exp Condition 3; Exp Condition 4; Exp Condition 5; Exp Condition 6; Exp Condition 7; Exp Condition 8
Behavioral: Buddy — Participants assigned to this condition will select a buddy of their choice (i.e. friend, co-worker, caregiver or family member) that is ≥ 18 years of age and willing to share their Fitbit data with the study team. The buddy will be mailed a Fitbit, share their Fitbit data with the study team, and be provided with access to, and instructions for, all of the study app modules the participant has access to for their assigned condition.
  The study app include a buddy module where the buddy and participant can view each other's progress. The buddy will be expected to attend a 15-30 minute group orientation call and listen to four 10-15 minute podcast (one every 3 weeks) during the first 24 weeks of the intervention. Each webinar will provide social support training and peer discussion of challenges and successes in providing BCS with MVPA support.
  Arms: Exp Condition 1; Exp Condition 11; Exp Condition 13; Exp Condition 15; Exp Condition 3; Exp Condition 5; Exp Condition 7; Exp Condition 9
Behavioral: General Mindfulness Training — Participants assigned to this condition will be instructed to watch 1 (1-2 mins), mindfulness education videos each week which lay the foundation for what mindfulness is and how it can be an important health behavior. Each week participants will also be asked to listen to general guided mindfulness audio files ≥5 days/ week. The length of recordings will gradually increase each week from 3-5 to 25-30 minutes. All videos and recording will be available via the study app.
  Arms: Exp Condition 1; Exp Condition 10; Exp Condition 13; Exp Condition 14; Exp Condition 2; Exp Condition 5; Exp Condition 6; Exp Condition 9
Behavioral: MVPA-Specific Mindfulness Training — Participants assigned to the MVPA-specific mindfulness training component will be instructed to watch 1-2 brief (1-2 minute), mindfulness education videos each week which lay the foundation for what mindfulness is and the importance of linking mindful awareness with MVPA. Each week participants will be provided access to MVPA-specific guided mindfulness audio files (e.g., 10-minute treadmill walking meditation, 20-minute bicycling meditation) that they will be asked to listen to during ≥3 MVPA sessions/week. The length and intensity of these audio files will correspond to their progression in the program. All videos and recordings will be accessed via the study app.
  Arms: Exp Condition 1; Exp Condition 11; Exp Condition 12; Exp Condition 13; Exp Condition 14; Exp Condition 2; Exp Condition 7; Exp Condition 8

SUMMARY:
The primary purpose of the present study is to apply MOST methodology to determine which types of social support and mindfulness training intervention components optimally increase MVPA adoption and maintenance in Breast Cancer Survivors (BCS) in a 24-week intervention with a 48-week follow-up. The researchers will also examine the effects of changes in MVPA on symptom burden, time spent in intensities of other activities (i.e. light and sedentary), and sleep quality and duration.

Aim 1: To identify which components from four mHealth components under consideration for inclusion meaningfully contribute to improvements in MVPA at 24 and 48 weeks.

Aim 2: To examine how changes in MVPA, as a result of the 4 components, may influence additional health behaviors and outcomes including: a) symptom burden (i.e. fatigue, depression, anxiety); b) time spent i n other activity intensities (i.e. light, sedentary time); and c) sleep duration and quality.

Aim 3: To examine potential mediators (i.e. adherence, psychosocial factors such as post-traumatic growth, self-compassion, self-efficacy, and goal-setting) and moderators (i.e., age, time since diagnosis) of the four intervention components on MVPA.

DETAILED DESCRIPTION:
The primary purpose of the present study is to apply MOST methodology to determine which types of social support and mindfulness training intervention components optimally increase MVPA adoption and maintenance in Breast Cancer Survivors (BCS) in a 24-week intervention with a 48-week follow-up. The researchers will also examine the effects of changes in MVPA on symptom burden, time spent in intensities of other activities (i.e. light and sedentary), and sleep quality and duration.

Aim 1: To identify which components from four mHealth components under consideration for inclusion meaningfully contribute to improvements in MVPA at 24 and 48 weeks.

Aim 2: To examine how changes in MVPA, as a result of the 4 components, may influence additional health behaviors and outcomes including: a) symptom burden (i.e. fatigue, depression, anxiety); b) time spent i n other activity intensities (i.e. light, sedentary time); and c) sleep duration and quality.

Aim 3: To examine potential mediators (i.e. adherence, psychosocial factors such as post-traumatic growth, self-compassion, self-efficacy, and goal-setting) and moderators (i.e., age, time since diagnosis) of the four intervention components on MVPA.

Research participants will be identified and recruited at Robert H. Lurie Cancer Center (RHLCC) at Northwestern University (NU). All BCS and Buddies will complete an initial 10-15 minute eligibility screening online, over the phone, or in-person. The study RA will obtain informed consent and HIPAA authorization from eligible participants according to IRB approved procedures.

Assessments. After informed consent completion, the NU study team will send participants an email with an individual, secure link to study questionnaires and notification that an ActiGraph accelerometer packet has been mailed. Participants will be asked to complete the questionnaire within 1 week of receipt. BCS will be provided with detailed written instructions for how to wear the ActiGraph.

Randomization and Study Orientation. After completing baseline assessments, BCS will be randomized to each group using computer-generated randomly permuted blocks. After randomization, the NU study team will send the participant an intervention packet which will include the Fitbit, Fitbit instructions, instructions and a QR code to download the study app, and instructions specific to each condition to which they are assigned. The participant will also be scheduled for an orientation phone or web call with study staff to go over the contents of the intervention packet and expectations of participation for each component in greater detail.

Intervention Components

Core Intervention (Fitbit + Study App). All participants will receive a low-resource self-monitoring intervention consisting of the Fitbit AltaHR (or similar) and the study self-monitoring app. Participants will be asked to download the Fitbit app and wear the Fitbit 24/7 throughout the 48-week study period. The core study app will support BCS to increase their MVPA. Participants will be provided with a weekly MVPA goal to build efficacy and ensure safe progression towards the overall goal of 150 minutes per week. Participants will be instructed to self-monitor progress towards these goals via feedback on Fitbit Alta HR and the daily, weekly and monthly progress information provided in the study app.

Buddy. Participants assigned to this condition will select a buddy of their choice (i.e. friend, co-worker, caregiver or family member) that is ≥ 18 years of age and willing to share their Fitbit data with the study team. The study team will reach out to the buddy via an email containing a description of the expectations of the buddy and a link to complete online screening. The buddy will be mailed a Fitbit, share their Fitbit data with the study team, and be provided with access to, and instructions for, all of the study app modules the participant has access to for their assigned condition. The buddy will be expected to attend a 15-minute group orientation call online and to listen to four 10-15 minute podcasts (one every 3 weeks) during the 24 week intervention. Each webinar will provide social support training and peer discussion of challenges and successes in providing BCS with MVPA support.

E-coaching. Participants assigned to this condition will receive a weekly scheduled text message from their coach. Text messages will focus on building self-efficacy and self-regulation skills, setting realistic outcome expectations, overcoming barriers, and problem-solving and will directly support the participant's engagement in the intervention. The coach will provide a brief overview of the participant's recent progress and goals, ask if they are having any barriers and help them troubleshoot and set specific goals for the next week. In addition to the scheduled messaging, participants will also be instructed to reach out to their coach with any questions or for additional assistance. The coach will respond within 24 hours (weekdays) to 48 hours (weekends), maximum.

General Mindfulness Training. Participants assigned to this condition will be instructed to watch 1 (1-2 mins), mindfulness education videos each week which lay the foundation for what mindfulness is and how it can be an important health behavior. Each week participants will also be asked to listen to general guided mindfulness audio files ≥5 days/ week. The length of recordings will gradually increase each week from 3-5 to 25-30 minutes. All videos and recording will be available via the study app.

MVPA-Specific Mindfulness Training. Participants assigned to the MVPA-specific mindfulness training component will be instructed to watch 1-2 brief (1-2 minute), mindfulness education videos each week which lay the foundation for what mindfulness is and the importance of linking mindful awareness with MVPA. Each week participants will be provided access to MVPA-specific guided mindfulness audio files (e.g., 10-minute treadmill walking meditation, 20-minute bicycling meditation) that they will be asked to listen to during ≥3 MVPA sessions/week. The length and intensity of these audio files will correspond to their progression in the program. All videos and recording will be accessed via the study app.

Follow-up. Participants will be instructed to maintain their MVPA during the 24-week follow-up period. They will have access to all materials to which they were assigned to less any direct contact from the study team.

ELIGIBILITY:
Inclusion Criteria:

For BCS

* Female, age 18 years or older
* Stage I-III breast cancer diagnosis within the past 5 years
* Diagnosis of cancer between 18-39 years and within the past 5 years
* ≥3 months post-completion of primary treatment (i.e., surgery, chemotherapy, and/or radiation); may still be undergoing endocrine or hormone therapies
* Self-report engagement in <60 min/week of MVPA
* Score of 0 on all positive statement(s) of the Physical Activity Readiness Questionnaire (PAR-Q)18 or willingness to obtain medical clearance from a primary care physician or oncologist
* Internet access and smartphone ownership
* Fluency in spoken and written English
* Willingness to find a buddy (someone who knows about their cancer and participation in this study and who is willing to participate by supporting them during the 24-week study), if assigned to that condition

For "Buddies"

* Friend, co-worker, caregiver or family member of a participating BCS
* Age 18 years or older
* Score of 0 on all positive statement(s) of the Physical Activity Readiness Questionnaire (PAR-Q)18 or willing to obtain medical clearance from a primary care physician
* Internet access and smartphone ownership
* Fluency in spoken and written English
* Willingness to share their Fitbit data with the study team

Exclusion Criteria:

* Absolute contraindications to exercise (i.e., acute myocardial infarction, severe orthopedic conditions), metastatic disease, or planned elective surgery
* Currently pregnant or plans to become pregnant
* Plans to move out of the United States in next 18 months
* Current enrollment in another dietary or physical activity trial
* Inability to provide informed consent
* Prisoners or other detained individuals

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-03-24 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Objective Physical Activity during the 48 week technology supported physical activity interventions in breast cancer survivors | 48 weeks
  Physical activity will be measured at baseline, 24 and 48 weeks.The ActiGraph accelerometer will be used. At each time point, participants will wear the device for 7 consecutive days during all waking hours, except when bathing or swimming. Each valid minute of wear time will be classified according to intensity (counts/min) using commonly accepted cut-points: sedentary (<100), light activity (100-2019) and moderate/vigorous physical activity (≥2020). Minutes of moderate and vigorous physical activity will be used to assess change.

SECONDARY OUTCOMES:
Anxiety in breast cancer survivors | 48 weeks
  Symptom burden of anxiety will be measured at baseline, 24 and 48 weeks using the PROMIS Item Bank v1.0 - Emotional Distress - Anxiety - Short Form 8a.
Depression in breast cancer survivors | 48 weeks
  Symptom burden of depression will be measured at baseline, 24 and 48 weeks using the PROMIS Item Bank v1.0 - Emotional Distress - Depression-Short Form 8a.
Fatigue in breast cancer survivors | 48 weeks
  Symptom burden of fatigue will be measured at baseline, 24 and 48 weeks using the PROMIS Item Bank v1.0 - Fatigue - Short Form 8a.
Physical Function in breast cancer survivors | 48 weeks
  Physical function will be measured at baseline, 24 and 48 weeks using the PROMIS Item Bank v. 1.0 - Physical Function - Short Form 20a.
Sleep Disturbance in breast cancer survivors | 48 weeks
  Symptom burden of sleep disturbance will be measured at baseline, 24 and 48 weeks using the PROMIS Item Bank v1.0 - Sleep Disturbance - Short Form 8a.
Sleep Impairment in breast cancer survivors | 48 weeks
  Symptom burden of sleep disturbance will be measured at baseline, 24 and 48 weeks using the PROMIS Item Bank v. 1.0 - Sleep-Related Impairment - Short Form 8a.
Applied Cognition Abilities in breast cancer survivors | 48 weeks
  Symptom burden on applied cognitive abilities will be measured at baseline, 24 and 48 weeks using the PROMIS v1.0-Applied Cognition-Abilities-Short Form 8a.
Emotional Support in breast cancer survivors | 48 weeks
  Symptom burden on emotional support will be measured at baseline, 24 and 48 weeks using the PROMIS Item Bank v2.0 - Emotional Support.
Self-Esteem in breast cancer survivors | 48 weeks
  Symptom burden on self-esteem will be measured at baseline, 24 and 48 weeks using the Rosenberg Self-Esteem Scale.
  This scale assesses global self-esteem and consists of 10-items asking participants to indicate their level of agreement/disagreement with each statement. Sample items include: "I feel that I'm a person of worth, at least on an equal basis with others;" and "I am able to things as well as most people." Participants respond on a 5-point Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree). The minimum value one can score is 10, and the maximum is 50. Higher scores indicate a better outcome.
Social support for exercise in breast cancer survivors | 48 weeks
  Social support for exercise will be measured at baseline, 24 and 48 weeks using the Social Support for Exercise Scale.
  This scale assesses support for physical activity received from the following categories: family, friends, and other cancer survivors. Statements are scored on a Likert scale of 1 (never) to 5 (very often) for each of the three categories, with higher scores representing better outcome. The minimum value one can score for each category is 10, and the maximum is 50. The minimum value of the total measure is 30, and the maximum is 150. An additional "does not apply" response option is provided on the measure.
Physical self-perception in breast cancer survivors | 48 weeks
  Physical Self-Perception will be measured at baseline, 24 and 48 weeks using the Physical Self-Perception Profile-Physical Self-worth Subscale.
  This instrument used to assess self-esteem relative to several domains of physical functioning in a hierarchical, multidimensional fashion. The instrument contains a general physical self-worth scale (PSW) which subsumes four more specific scales of perceived sport competence (SPORT), physical condition (COND), attractive body (BODY), and strength (STRENGTH), with six items per scale. Participants indicated on a four-point scale the degree to which each item is characteristic or true of them. Responses range from 1 (not at all true) to 4 (completely true), with higher scores representing better outcome. The minimum value one can score is 6, and the maximum is 24.
Enjoyment of Physical Activity in young adult cancer survivors | 48 weeks
  Enjoyment of Physical Activity will be measured at baseline, 24 and 48 weeks using the Physical Activity Enjoyment Scale.
  This 18-item scale assesses enjoyment for physical activity by asking participants to rate "how you feel at the moment about the physical activity you have been doing" using a 7 point bipolar Likert scale, from 1 (I enjoy it) to 7 (I hate it). Eleven items are negatively worded and seven items are positively worded. After reverse scoring the 11 negatively worded items, an overall enjoyment for physical activity score is determined by summing the items, with a value range of 18-126 being possible. Higher scores indicate higher enjoyment, better outcome.
Leisure Time Physical Activity in breast cancer survivors | 48 weeks
  Leisure time physical activity will be measured at baseline, 24 and 48 weeks using the Godin Leisure Time Exercise Questionnaire Physical Activity.
  This is a measure of self-reported physical activity participation. Participants report "times per week" they participate in strenuous (e.g., jogging), moderate (e.g., fast walking), and mild (e.g., easy walking) exercise over the past 7 days and the "average duration each time you exercised (in minutes)" for each of the three activity categories. Weekly minutes of total, light, moderate, and vigorous activity are calculated by multiplying the frequency and time of each activity. This value is divided by 7 to obtain daily averages. The minimum value one can score is 0, and the maximum depends on the number of self-reported minutes of physical activity. Higher scores indicate better outcome.
Confidence in ability to be regularly active in breast cancer survivors | 48 weeks
  Confidence in ability to be regularly active will be measured at baseline, 24 and 48 weeks using the Exercise Self-Efficacy (EXSE).
  This short form assesses the participants' beliefs in their ability to be regularly active "for the next 12 weeks" on a scale from 0% (not at all confident) to 100% (completely confident), with higher scores representing better outcome.
Confidence in ability to be regularly active despite common barriers in breast cancer survivors | 48 weeks
  Confidence in ability to be regularly active despite common barriers will be measured at baseline, 24 and 48 weeks using the Barries Self-Efficacy (BARSE).
  This scale assesses the beliefs in ability to be regularly active despite common barriers "for the next 12 weeks" on a scale from 0% (not at all confident) to 100% (completely confident), with higher scores representing better outcome.
Exercise goal setting in breast cancer survivors | 48 weeks
  Exercise goal setting in breast cancer survivors will be measured at baseline, 24 and 48 weeks using the Exercise Goal Setting Scale.
  This scale assesses exercise goal setting behaviors on a scale from 1 (does not describe) to 5 (describes completely), with higher scores representing better outcome.
Sitting time in breast cancer survivors | 48 weeks
  Sitting time in breast cancer survivors will be assessed at baseline, 24 and 48 weeks using the Sitting Time Questionnaire.
  This questionnaire assesses the amount of hours and minutes spent sitting during weekdays and weekends, with lower scores representing better outcome.
Outcome expectations for exercise in breast cancer survivors | 48 weeks
  Outcome expectations for exercise in breast cancer survivors will be assessed at baseline, 24 and 48 weeks using the Outcome Expectations for Exercise_MOEES.
  This scale assesses the beliefs and expectations about the benefits of regular exercise and physical activity on a scale from 1 (strongly disagree) to 5 (strongly agree), with higher scores representing better outcome.
Mindful Awareness in breast cancer survivors | 48 weeks
  Mindful awareness of distressing thoughts and images will be measured at baseline, 24 and 48 weeks using the Southampton Mindfulness Questionnaire (SMQ).
  This 16-item scale measures mindful awareness during distressing thoughts and images. Using a 7-point Likert scale (0=strongly disagree to 6=strongly agree), items reflect the following subscales: mindful observation (4 items), letting go (4 items), non- aversion (4 items), and non-judgment (4 items). The minimum value one can score on any of the subscales is 0, and the maximum is 24. The minimum value of the total measure is 0, and the maximum is 96. The higher scores represent better outcome.
Mindful self-compassion in breast cancer survivors | 48 weeks
  Mindful self-compassion will be measured at baseline, 24 and 48 weeks using the Self-Compassion Short Form.
  This short form is a 12-item scale measuring items related to self-kindness, self-judgment, and common humanity. Statements on the Self-Compassion Scale are scored on a Likert scale of 1 (almost never) to 5(almost always). To calculate an overall compassion score - Items representing uncompassionate responses to inadequacy or suffering (the self-judgment, isolation, and over-identification subscales) are reverse-coded only when calculating the overall compassion score. In this way, higher scores represent a lower frequency of these responses.
Post-traumatic growth in breast cancer survivors | 48 weeks
  Post-traumatic growth will be measured at baseline, 24 and 48 weeks using the Post-traumatic Growth Inventory.
  This 21-item self-report scale assesses growth or benefits after a specific traumatic life event. The Post Traumatic Growth Inventory (PTGI) is scored by adding all the responses, with higher scores representing better outcome.
Implementation feasibility measured by enrollment rate | 48 weeks
  This indicator of implementation feasibility for the interventions delivered is defined by the overall enrollment rate being >/= 70% (e.g., total number of individuals enrolled/total number approached). Enrollment rate will be tracked continuously during the 48 week study.
Implementation feasibility measured by retention rate | 48 weeks
  This indicator of implementation feasibility for the interventions delivered is defined by the retention rate being >/= 70% (e.g., total number of participants who drop out/ total number randomized). Retention rate will be tracked continuously during the 48 weeks of the study and significant differences between the study interventions in the number of participant withdrawals will be tracked.
Adherence to the study app + Fitbit by breast cancer survivors | 48 weeks
  Adherence to the study app + Fitbit will be monitored and usage tracked continuously during the 48 week study.
  Objective data include Fitbit wear time, number of times app is opened each week, time spent in app each time it is opened, and for participants who receive each component, usage of general and moderate to vigorous intensity physical activity specific mindfulness videos (i.e. whether clicked, how many times and for how long), number of e-coaching exchanges, number of buddy training webinars attended, and number of buddy interactions in the app.
Acceptability of the technology supported physical activity interventions as measured by a post-intervention evaluation survey | 48 weeks
  Acceptability will be measured using a brief, Likert-type survey assessing participant enjoyment, satisfaction, perceived benefit, and ease of use. Acceptability is defined as >/= 70% of survey responses in affirmation of this.
Change in body mass index in breast cancer survivors | 48 weeks
  Change in body mass index in breast cancer survivors will be assessed at baseline, 24 and 48 weeks using the Health History Questionnaire, a local questionnaire developed by the study researchers.
  Participants will report on the following: height and most recent weight. BMI will be calculated. Significant change will be indicated by p<.05 on reported health behaviors between baseline and follow up time points between study interventions.
Change in health behaviors in breast cancer survivors | 48 weeks
  Change in health behaviors in breast cancer survivors will be assessed at baseline, 24 and 48 weeks using the Health History Questionnaire, a local questionnaire developed by the study researchers.
  Participants will report on the following: weekly leisure-time physical activities; weekly consumption of fruits, vegetables, fast food/snacks, caffeine, carbonated beverages; cigarette and alcohol use. Unhealthy behaviors will be reverse scored. Higher scores represent better outcome. Significant change will be indicated by p<.05 on reported health behaviors between baseline and follow up time points between study interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan M Phillips, PhD, MPH, Principal Investigator — Northwestern University; David E Victorson, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller KD, Nogueira L, Mariotto AB, Rowland JH, Yabroff KR, Alfano CM, Jemal A, Kramer JL, Siegel RL. Cancer treatment and survivorship statistics, 2019. CA Cancer J Clin. 2019 Sep;69(5):363-385. doi: 10.3322/caac.21565. Epub 2019 Jun 11. PMID 31184787
- [Background] Ibrahim EM, Al-Homaidh A. Physical activity and survival after breast cancer diagnosis: meta-analysis of published studies. Med Oncol. 2011 Sep;28(3):753-65. doi: 10.1007/s12032-010-9536-x. Epub 2010 Apr 22. PMID 20411366
- [Background] McNeely ML, Campbell KL, Rowe BH, Klassen TP, Mackey JR, Courneya KS. Effects of exercise on breast cancer patients and survivors: a systematic review and meta-analysis. CMAJ. 2006 Jul 4;175(1):34-41. doi: 10.1503/cmaj.051073. PMID 16818906
- [Background] Speck RM, Courneya KS, Masse LC, Duval S, Schmitz KH. An update of controlled physical activity trials in cancer survivors: a systematic review and meta-analysis. J Cancer Surviv. 2010 Jun;4(2):87-100. doi: 10.1007/s11764-009-0110-5. Epub 2010 Jan 6. PMID 20052559
- [Background] Ballard-Barbash R, Friedenreich CM, Courneya KS, Siddiqi SM, McTiernan A, Alfano CM. Physical activity, biomarkers, and disease outcomes in cancer survivors: a systematic review. J Natl Cancer Inst. 2012 Jun 6;104(11):815-40. doi: 10.1093/jnci/djs207. Epub 2012 May 8. PMID 22570317
- [Background] Arem H, Mama SK, Duan X, Rowland JH, Bellizzi KM, Ehlers DK. Prevalence of Healthy Behaviors among Cancer Survivors in the United States: How Far Have We Come? Cancer Epidemiol Biomarkers Prev. 2020 Jun;29(6):1179-1187. doi: 10.1158/1055-9965.EPI-19-1318. Epub 2020 May 14. PMID 32409489
- [Background] Thraen-Borowski KM, Gennuso KP, Cadmus-Bertram L. Accelerometer-derived physical activity and sedentary time by cancer type in the United States. PLoS One. 2017 Aug 14;12(8):e0182554. doi: 10.1371/journal.pone.0182554. eCollection 2017. PMID 28806753
- [Background] Devoogdt N, Van Kampen M, Geraerts I, Coremans T, Fieuws S, Lefevre J, Philippaerts R, Truijen S, Neven P, Christiaens MR. Physical activity levels after treatment for breast cancer: one-year follow-up. Breast Cancer Res Treat. 2010 Sep;123(2):417-25. doi: 10.1007/s10549-010-0997-6. Epub 2010 Jun 27. PMID 20582717
- [Background] Charlier C, Van Hoof E, Pauwels E, Lechner L, Spittaels H, De Bourdeaudhuij I. The contribution of general and cancer-related variables in explaining physical activity in a breast cancer population 3 weeks to 6 months post-treatment. Psychooncology. 2013 Jan;22(1):203-11. doi: 10.1002/pon.2079. Epub 2011 Oct 5. PMID 22052746
- [Background] Irwin ML, Crumley D, McTiernan A, Bernstein L, Baumgartner R, Gilliland FD, Kriska A, Ballard-Barbash R. Physical activity levels before and after a diagnosis of breast carcinoma: the Health, Eating, Activity, and Lifestyle (HEAL) study. Cancer. 2003 Apr 1;97(7):1746-57. doi: 10.1002/cncr.11227. PMID 12655532
- [Background] Phillips SM, McAuley E. Social cognitive influences on physical activity participation in long-term breast cancer survivors. Psychooncology. 2013 Apr;22(4):783-91. doi: 10.1002/pon.3074. Epub 2012 Mar 26. PMID 22451113
- [Background] Thorsen L, Courneya KS, Stevinson C, Fossa SD. A systematic review of physical activity in prostate cancer survivors: outcomes, prevalence, and determinants. Support Care Cancer. 2008 Sep;16(9):987-97. doi: 10.1007/s00520-008-0411-7. Epub 2008 Feb 15. PMID 18274783
- [Background] Stevinson C, Tonkin K, Capstick V, Schepansky A, Ladha AB, Valance JK, Faught W, Steed H, Courneya KS. A population-based study of the determinants of physical activity in ovarian cancer survivors. J Phys Act Health. 2009 May;6(3):339-46. doi: 10.1123/jpah.6.3.339. PMID 19564663
- [Background] Kampshoff CS, Jansen F, van Mechelen W, May AM, Brug J, Chinapaw MJ, Buffart LM. Determinants of exercise adherence and maintenance among cancer survivors: a systematic review. Int J Behav Nutr Phys Act. 2014 Jul 2;11:80. doi: 10.1186/1479-5868-11-80. PMID 24989069
- [Background] Valle CG, Tate DF. Engagement of young adult cancer survivors within a Facebook-based physical activity intervention. Transl Behav Med. 2017 Dec;7(4):667-679. doi: 10.1007/s13142-017-0483-3. PMID 28374211
- [Background] Schneider J, Malinowski P, Watson PM, Lattimore P. The role of mindfulness in physical activity: a systematic review. Obes Rev. 2019 Mar;20(3):448-463. doi: 10.1111/obr.12795. Epub 2018 Nov 23. PMID 30468299
- [Background] Rabin C, Pinto B, Fava J. Randomized Trial of a Physical Activity and Meditation Intervention for Young Adult Cancer Survivors. J Adolesc Young Adult Oncol. 2016 Mar;5(1):41-7. doi: 10.1089/jayao.2015.0033. Epub 2015 Oct 15. PMID 26812450
- [Background] Courneya KS, Rogers LQ, Campbell KL, Vallance JK, Friedenreich CM. Top 10 research questions related to physical activity and cancer survivorship. Res Q Exerc Sport. 2015 Jun;86(2):107-16. doi: 10.1080/02701367.2015.991265. Epub 2015 Jan 28. PMID 25629322
- [Background] Hedeker D, Gibbons RD, Waternaux C. Sample size estimation for longitudinal designs with attrition: comparing time-related contrasts between two groups. Journal of Educational and Behavioral Statistics. 1999;24(1):70-93.
- [Background] Buchholz SW, Wilbur J, Ingram D, Fogg L. Physical activity text messaging interventions in adults: a systematic review. Worldviews Evid Based Nurs. 2013 Aug;10(3):163-73. doi: 10.1111/wvn.12002. Epub 2013 Jun 7. PMID 23746267
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] Welk GJ, McClain JJ, Eisenmann JC, Wickel EE. Field validation of the MTI Actigraph and BodyMedia armband monitor using the IDEEA monitor. Obesity (Silver Spring). 2007 Apr;15(4):918-28. doi: 10.1038/oby.2007.624. PMID 17426327
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Garcia SF, Cella D, Clauser SB, Flynn KE, Lad T, Lai JS, Reeve BB, Smith AW, Stone AA, Weinfurt K. Standardizing patient-reported outcomes assessment in cancer clinical trials: a patient-reported outcomes measurement information system initiative. J Clin Oncol. 2007 Nov 10;25(32):5106-12. doi: 10.1200/JCO.2007.12.2341. PMID 17991929
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Lai J-S, Cella D, Choi S, Teresi JA, Hays RD, Stone AA. Developing a fatigue item bank for the Patient-Reported Outcomes Measurement Information System (PROMIS FIB version 1). Presented at the Meeting of the Survey Methods in Multicultural, Multinational, and Multiregional Contexts (3MC), Berlin, Germany. 2008.
- [Background] Buysse DJ, Yu L, Moul DE, Germain A, Stover A, Dodds NE, Johnston KL, Shablesky-Cade MA, Pilkonis PA. Development and validation of patient-reported outcome measures for sleep disturbance and sleep-related impairments. Sleep. 2010 Jun;33(6):781-92. doi: 10.1093/sleep/33.6.781. PMID 20550019
- [Background] Chadwick P, Hember M, Symes J, Peters E, Kuipers E, Dagnan D. Responding mindfully to unpleasant thoughts and images: reliability and validity of the Southampton mindfulness questionnaire (SMQ). Br J Clin Psychol. 2008 Nov;47(Pt 4):451-5. doi: 10.1348/014466508X314891. Epub 2008 Jun 20. PMID 18573227
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Tedeschi RG, Calhoun LG. The Posttraumatic Growth Inventory: measuring the positive legacy of trauma. J Trauma Stress. 1996 Jul;9(3):455-71. doi: 10.1007/BF02103658. PMID 8827649
- [Background] McAuley E. Self-efficacy and the maintenance of exercise participation in older adults. J Behav Med. 1993 Feb;16(1):103-13. doi: 10.1007/BF00844757. PMID 8433355
- [Background] Wojcicki TR, White SM, McAuley E. Assessing outcome expectations in older adults: the multidimensional outcome expectations for exercise scale. J Gerontol B Psychol Sci Soc Sci. 2009 Jan;64(1):33-40. doi: 10.1093/geronb/gbn032. Epub 2009 Jan 29. PMID 19181688
- [Background] Rovniak LS, Anderson ES, Winett RA, Stephens RS. Social cognitive determinants of physical activity in young adults: a prospective structural equation analysis. Ann Behav Med. 2002 Spring;24(2):149-56. doi: 10.1207/S15324796ABM2402_12. PMID 12054320
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Rosenberg, M. Society and the adolescent self-image. Princeton, NJ: Princeton University Press.1965.
- [Background] Fox, K.R., & Corbin, C.B. The physical self-perception profile: Development and preliminary validation. Journal of Sport & Exercise Psychology, 11, 408-430 1989.
- [Background] Kendzierski D, DeCarlo KJ. Physical Activity Enjoyment Scale: Two validation studies. Journal of Sport & Exercise Psychology. 1991.
- [Background] Hedeker DR, Gibbons RD. Longitudinal Data Analysis. Hoboken, N.J.: Wiley-Interscience; 2006.
- [Background] Collins LM, Baker TB, Mermelstein RJ, Piper ME, Jorenby DE, Smith SS, Christiansen BA, Schlam TR, Cook JW, Fiore MC. The multiphase optimization strategy for engineering effective tobacco use interventions. Ann Behav Med. 2011 Apr;41(2):208-26. doi: 10.1007/s12160-010-9253-x. PMID 21132416
- [Background] Collins LM, Murphy SA, Nair VN, Strecher VJ. A strategy for optimizing and evaluating behavioral interventions. Ann Behav Med. 2005 Aug;30(1):65-73. doi: 10.1207/s15324796abm3001_8. PMID 16097907
- [Background] Pinheiro JC, Bates DM. Approximations to the log-likelihood function in the nonlinear mixed-effects model. Journal of Computational and Graphical Statistics. 1995;4(1):12-35.
- [Background] Krull JL, MacKinnon DP. Multilevel Modeling of Individual and Group Level Mediated Effects. Multivariate Behav Res. 2001 Apr 1;36(2):249-77. doi: 10.1207/S15327906MBR3602_06. PMID 26822111
- [Background] DiCiccio TJ, Efron B. Bootstrap confidence intervals. Statistical science. 1996:189-212.
- [Background] Hankin VV, D.; Polster, R. . Maximizing Acceptance and Enrollment in MBSR Randomized Controlled Trials with Older Men Diagnosed with Cancer. . Poster presented to the 8th Annual International Scientific Conference of Mindfulness in Medicine, Health Care, and Society Worcester, MA. 2010.
- [Background] Victorson D, Du H, Hankin V, et al. Mindfulness-based stress reduction decreases fear of progression over time for men with prostate cancer on active surveillance: results from a randomized clinical trial. J Urol. 2012;187(4S):384.
- [Background] Victorson D, Hankin V, Burns J, Weiland R, Maletich C, Sufrin N, Schuette S, Gutierrez B, Brendler C. Feasibility, acceptability and preliminary psychological benefits of mindfulness meditation training in a sample of men diagnosed with prostate cancer on active surveillance: results from a randomized controlled pilot trial. Psychooncology. 2017 Aug;26(8):1155-1163. doi: 10.1002/pon.4135. Epub 2016 May 3. PMID 27145355
- [Background] Victorson D, Maletich C, Gutierrez B, Schuette S, Morgan T, Kutikov A, Kundu S, Eggener S, Brendler C. Description of a new national cancer institute funded randomized controlled trial
- [Background] Victorson D, Garland, E, Hanley, A, Greco, C. Is mindfulness immeasurable? Discovery and dialogue of conceptual, practical, scientific, and experiential solutions. Glob Adv Health Med. 2018 7(1160):13.
- [Background] Victorson D, Maletich, C, Sufrin, N, Schuette, S, Gutierrez, B, Cordero, E, Johnson, C, Stencel, D, Bakosh, L, Ring, M. Development of a New Clinical Mindfulness Research Tool to Enhance, Deliver and Streamline Online Mindfulness Interventions. J Altern Complement Med. 2016;0(0):A21.
- [Derived] Wolter M, Reading JM, Solk P, Starikovsky J, Hasanaj K, Wang SD, Siddique J, Horowitz B, Spring B, Carden LB, Fox R, Sauer C, Freeman H, Frey J, Victorson D, Phillips SM. Optimizing a mHealth physical activity intervention with mindful awareness lessons in breast cancer survivors: Fit2ThriveMIND protocol. Contemp Clin Trials. 2025 Sep;156:108038. doi: 10.1016/j.cct.2025.108038. Epub 2025 Jul 31. PMID 40752821